CLINICAL TRIAL: NCT03739775
Title: Circulating Tumor DNA for the Early Detection of HPV-positive Pelvic Cancer Relapses
Brief Title: Circulating Tumor DNA for the Early Detection of HPV-positive Pelvic Cancer Relapses (CIRCA-HPV)
Acronym: CIRCA-HPV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2017-01
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: HPV Positive Pelvic Cancer
Keywords: HPV positive pelvic cancer; Circulating tumor biomarker
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sampling (Other)
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Patients will have a blood draw at each visit to the hospital and at least 6 months (+/- 1 month) intervals.

SUMMARY:
ctDNA detection in patients with previously treated, HPV-induced, stage II or III invasive pelvic cancer and who are currently in post-treatment follow-up.

DETAILED DESCRIPTION:
Patients with previously treated, HPV-induced, stage II or III invasive pelvic cancer and who are currently in post-treatment follow-up will be included.

These patients will be followed up during 30 months (2.5 years) (if no relapse occurred before) with ctDNA detection performed at each hospital visit. At each visit, clinical, biological (squamous cell carcinoma (SCC) serum marker will be done systematically) and radiological/pathology (if any) results will be prospectively collected in the study.

For the patients who have a relapse or new HPV-induced invasive cancer before 30 months, the follow-up will be discontinued at the date of the relapse.

For the patients who will have completed their follow-up for the study (2.5 years) with no relapse or new HPV-induced invasive cancer, they will be followed up for 6 months (+ 14 days), to collect any late relapse (if any). None specific study procedure will be performed during this period.

ELIGIBILITY:
Inclusion Criteria:

1. 1) Patient curatively treated within the past 3 years for:

   * a HPV-induced stage Ib3, Ic, II or III cervix cancer
   * a HPV-induced stage II or III anal canal, vagina, vulva or penis cancer
2. Patient with no evidence of any invasive tumor at inclusion (clinical and, if any, radiological exams).
3. Age ≥ 18 years
4. Availability of HPV genotyping of the treated cancer and/or archived tumor tissue available.
5. Patient who a follow-up visit is scheduled in the including center at least twice a year.
6. Patient being affiliated to the French social security.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patient presenting with active invasive tumor masses (e.g. stage IV cancer).
2. Patient deprived from ability to decide on her own or placed under the authority of a tutor.
3. Patient unable to have a regular follow up for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of plasma circulating tumor DNA detection as a test to detect any (local or distant) relapse in patients who have been curatively treated for HPV-induced invasive pelvic cancer (cervix, anal canal, vagina, vulva, penis). | up to 36 months
  Sensitivity= % of patients with number of copies/ml of ctDNA > threshold among those who experience a relapse within 6 months (+14 days) after the blood draw.
Specificity of plasma circulating tumor DNA detection as a test to detect any (local or distant) relapse in patients who have been curatively treated for HPV-induced invasive pelvic cancer (cervix, anal canal, vagina, vulva, penis). | up to 36 months
  Specificity= % of patients with number of copies/ml of ctDNA < threshold among those who don't experience a relapse within the 6 months after the blood draw (+14 days)

SECONDARY OUTCOMES:
Positive predictive values of ctDNA. | up to 36 months
  Positive Predictive Value= Probability of being diagnosed with a relapse within 6 months (+14 days) after positive testing (number of copies of ctDNA in the plasma > threshold).
Negative predictive values of ctDNA. | up to 36 months
  Negative Predictive Value= Probability of being relapse-free during the 6 months (+14 days) after negative testing (number of copies of ctDNA in the plasma < threshold).

CONTACTS AND LOCATIONS:
Overall Officials: François-Clément BIDARD, PhD, Principal Investigator — Institut Curie Paris
Locations (5):
- France (5):
  - CHU de Besançon, Besançon
  - Institut Curie - Paris, Paris
  - Hôpital Tenon, Paris
  - CHU Pontchaillou, Rennes
  - Institut Curie - Saint-Cloud, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).